CLINICAL TRIAL: NCT06587347
Title: Effects of Tirofiban on Early Neurological Deterioration After Intravenous Thrombolysis in Patients with Acute Ischemic Stroke: an Open-label, Multicenter, Randomized Controlled Trial
Brief Title: Tirofiban for the Prevention of Early Neurological Deterioration After Intravenous Thrombolysis in Acute Ischemic Stroke
Acronym: TREND-2
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TREND-2
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: Acute Stroke; Ischemic Stroke, Acute; Cerebral Infarction
Keywords: Acute ischemic stroke; Neurological deterioration; Stroke progression; intravenous thrombolysis; Antiplatelet therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebral Infarction | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirofiban Group (Experimental): Patients will receive tirofiban in the first 24 hours after intravenous thrombolysis, then bridge to oral antiplatelet therapy.
  Interventions: Drug: Tirofiban Hydrochloride
- Control group (Active Comparator): Aspirin, clopidogrel, or other antiplatelet drugs will be used in principle after 24 hours of thrombolytic therapy or until the primary outcome occurs.
  Interventions: Drug: Standard medical treatment (SMT)

INTERVENTIONS:
Drug: Tirofiban Hydrochloride — Tirofiban will use a loading dose, 0.4 μg/kg/min × 30 minutes, then 0.1μg/kg/min infusion until 24 hours after Intravenous thrombolytic therapy, or use a loading dose, 25 μg/kg, administrated within 3 minutes, then 0.15μg/kg/min infusion until 24 hours after Intravenous thrombolytic therapy.
  Arms: Tirofiban Group
Drug: Standard medical treatment (SMT) — Patients will receive standard antiplatelet therapy.
  Arms: Control group

SUMMARY:
A prospective, multicenter, randomized, controlled, open-label, blinded endpoint trial to evaluate the safety and efficacy of intravenous administration of tirofiban for preventing early neurological deterioration after intravenous thrombolysis in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Intravenous thrombolysis with recombinant tissue plasminogen activator (rt-PA), administered within 4.5 hours of symptom onset, remains the standard treatment strategy for acute ischemic stroke. However, approximately 6-40% of patients experienced early neurological deterioration following intravenous thrombolysis, among which more than 70% resulted from ischemic events, with 20-34% due to early re-occlusion of the recanalized artery. Augmented platelet activation, triggered by the activated coagulation cascade and endothelial injury during rt-PA administration, is recognized as one of the primary reasons for ischemic events after intravenous thrombolysis. Early antiplatelet therapy following rt-PA effectively reduces neurological deterioration and improves functional outcomes. However, the current guidelines recommend that antiplatelet therapy should be initiated 24 hours after intravenous thrombolysis due to the potential risk of intracerebral hemorrhage.

Tirofiban, a glycoprotein (GP) IIb/IIIa receptor inhibitor renowned for its rapid action, high selectivity, and short half-life, has been found to exert a remarkable antiplatelet effect by effectively blocking the terminal pathway that triggers platelet aggregation. One recent randomized trial found that among patients with acute non-cardioembolic ischemic stroke who presented within 24 hours of symptom onset, intravenous tirofiban resulted in a lower likelihood of early neurological deterioration than oral aspirin, without increasing the risk of intracranial hemorrhage or systematic bleeding. Another randomized trial found that treatment with intravenous tirofiban administration was safe and significantly improved 3-month functional outcomes in patients who experienced early neurological deterioration or no improvement within 24 hours of intravenous thrombolysis, compared with aspirin. Furthermore, our previous study found that early administration of tirofiban in patients with early neurological deterioration within the first 24 hours of intravenous thrombolysis did not increase the risk of symptomatic intracerebral hemorrhage, any intracerebral hemorrhage, or mortality. In contrast, it was associated with neurological improvement at 3 months. However, whether early administration of tirofiban can safely and effectively prevent neurological deterioration in patients with acute ischemic stroke treated with intravenous thrombolysis within 24 hours remains unclear, while the subset of patients who may benefit from early antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Acute ischemic stroke treated with intravenous thrombolysis with alteplase or tenecteplase within 4.5 hours of onset or time last known well and can receive the study drug treatment within 3 hours of initiating intravenous thrombolysis.
3. Residual NIHSS score ≥ 5 points at randomization (at least 1 hour after intravenous thrombolytic therapy).
4. Post-thrombolysis imaging shows that the offending artery is consistent with moderate or severe intracranial atherosclerotic stenosis (within 50%~99%)
5. Informed consent obtained from patients or their acceptable surrogates.

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by imaging post-thrombolysis.
2. Stroke caused by other determined causes, including moyamoya disease, artery dissection, arteritis, etc.
3. Scheduled for or received endovascular treatment after onset.
4. Definite or suspected cardioembolic stroke.
5. Definite anticipation of developing indications for anticoagulant therapy during the study period (e.g., atrial fibrillation, mechanical heart valve, deep vein thrombosis, pulmonary embolism, antiphospholipid syndrome, hypercoagulable state).
6. Use of antiplatelet or anticoagulant therapy within one week pre-stroke.
7. Pre-stroke mRS score ≥ 2.
8. Severe consciousness disturbance with NIHSS item 1a (level of consciousness) >1 point at randomization.
9. History of tirofiban allergy or its solvents.
10. History of platelet count < 100 × 109/L caused by tirofiban.
11. Major surgical operation within 6 weeks.
12. Major systemic hemorrhage within 30 days;
13. Determined coagulation disorders, platelet dysfunction, or platelet count < 100*109/L.
14. Currently pregnant or lactating;
15. Uncontrolled hypertension with systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg.
16. Acute pericarditis or hemorrhagic retinopathy.
17. Presence of malignant tumors, chronic hemodialysis, severe renal insufficiency (GFR < 30 ml/min or serum Cr > 220 μmol/L (2.5 mg/dl)), severe hepatic insufficiency (serum ALT > 2 times the upper limit of normal, or serum AST > 2 times the upper limit of normal), severe heart failure (NYHA class III or IV).
18. Severe non-cardiovascular complications with an expected survival of less than 6 months.
19. Unavailability for follow-up.
20. Presence of dementia, psychiatric disorders, or other known neurological conditions that complicate follow-up.
21. Participated in this study in the past.
22. Current participation in another therapeutic study with ongoing treatment and follow-up.
23. Other conditions that are not suitable for participation in this study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing neurological deterioration within 24 hours after intravenous thrombolysis. | Within 24 hours after intravenous thombolysis.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale ranging from 0-42. A higher score means more severe stroke symptoms. Neurological deterioration is defined as an increase in NIHSS by ≥ 4 points compared to the lowest NIHSS.

SECONDARY OUTCOMES:
Change of the NIHSS | 7 days or discharge after intravenous thrombolytic therapy
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
The proportion of patients with a modified Rankin scale (mRS) score of 0-1 at 30-day follow up. | 30 days after stroke
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
The proportion of patients with a modified Rankin scale (mRS) score of 0-1 at 90-day follow up. | 90 days after stroke
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
The proportion of patients with a modified Rankin scale (mRS) score of 0-2 at 30-day follow up. | 30 days after stroke
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
The proportion of patients with a modified Rankin scale (mRS) score of 0-2 at 90-day follow up. | 90 days after stroke
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
Distribution of modified Rankin Scale (mRS) scores at 90 day. | 90 days after stroke
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
Incidence of symptomatic intracranial hemorrhage within 24 hours of intervention. | Within 24 hours of intervention
  Symptomatic intracranial hemorrhage is defined as the demonstration of hemorrhage within brain parenchyma on head imaging leading to an increase of at least 4 points in the NIHSS score, according to the criteria of the European Cooperative Acute Stroke Study III (ECASS III).
Incidence of any intracranial hemorrhage within 24 hours of intervention. | Within 24 hours of intervention
  Any intracranial hemorrhage is defined as the demonstration of hemorrhage within brain parenchyma on head imaging, according to the criteria of the ECASS III.
Incidence of systemic hemorrhage within 90 days after stroke. | Within 90 days after stroke.
  The incidence of systemic hemorrhage at any time from randomization through day 90, according to the criteria of the GUSTO.
Incidence of recurrent stroke or other vascular events within 90 days after stroke. | Within 90 days after stroke.
  The incidence of recurrent stroke or other vascular events (including hemorrhagic and ischemic stroke, myocardial infarction, and cardiovascular death) within 90 days of randomization.
All-cause death within 90 days after stroke. | Within 90 days after stroke.
  The incidence of death events at any time from randomization through day 90.
Incidence of Adverse Events/Serious Adverse Events within 90 days after stroke. | Within 90 days after stroke.
  The incidence of other adverse events and serious adverse events at any time from randomization through day 90.
Proportion of patients experiencing neurological deterioration (an increase in NIHSS by ≥ 2 points compared to the lowest NIHSS) within 24 hours after intravenous thrombolysis. | Within 24 hours of intravenous thrombolysis.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Proportion of patients experiencing neurological deterioration (an increase in NIHSS by ≥ 4 points compared to the lowest NIHSS) within 48 hours after intravenous thrombolysis. | Within 48 hours after intravenous thrombolysis.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Proportion of patients experiencing (an increase in NIHSS by ≥ 4 points compared to the lowest NIHSS) within 72 hours after intravenous thrombolysis. | Within 72 hours after intravenous thrombolysis.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Proportion of patients experiencing neurological deterioration (an increase in NIHSS by ≥ 4 points compared to the lowest NIHSS) within 7 days after intravenous thrombolysis. | Within 7 days after intravenous thrombolysis.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Proportion of patients with a decrease in NIHSS by ≥ 2 points compared to NIHSS at randomization. | 24 hours after intravenous thrombolysis.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.

OTHER OUTCOMES:
Biomarkers levels of groups | Within 24 hours of intervention
  The biomarkers include CLEC2, CD62P, TXB2, 6-k-PGFla, EETs, 20-HETE, BCAA, ALDH2

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao W, Li S, Li C, Wu C, Wang J, Xing L, Wan Y, Qin J, Xu Y, Wang R, Wen C, Wang A, Liu L, Wang J, Song H, Feng W, Ma Q, Ji X; TREND Investigators. Effects of Tirofiban on Neurological Deterioration in Patients With Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2024 Jun 1;81(6):594-602. doi: 10.1001/jamaneurol.2024.0868. PMID 38648030
- [Background] Zi W, Song J, Kong W, Huang J, Guo C, He W, Yu Y, Zhang B, Geng W, Tan X, Tian Y, Liu Z, Cao M, Cheng D, Li B, Huang W, Liu J, Wang P, Yu Z, Liang H, Yang S, Tang M, Liu W, Huang X, Liu S, Tang Y, Wu Y, Yao L, Shi Z, He P, Zhao H, Chen Z, Luo J, Wan Y, Shi Q, Wang M, Yang D, Chen X, Huang F, Mu J, Li H, Li Z, Zheng J, Xie S, Cai T, Peng Y, Xie W, Qiu Z, Liu C, Yue C, Li L, Tian Y, Yang D, Miao J, Yang J, Hu J, Nogueira RG, Wang D, Saver JL, Li F, Yang Q; RESCUE BT2 Investigators. Tirofiban for Stroke without Large or Medium-Sized Vessel Occlusion. N Engl J Med. 2023 Jun 1;388(22):2025-2036. doi: 10.1056/NEJMoa2214299. PMID 37256974
- [Background] Wu C, Sun C, Wang L, Lian Y, Xie N, Huang S, Zhao W, Ren M, Wu D, Ding J, Song H, Wang Y, Ma Q, Ji X. Low-Dose Tirofiban Treatment Improves Neurological Deterioration Outcome After Intravenous Thrombolysis. Stroke. 2019 Dec;50(12):3481-3487. doi: 10.1161/STROKEAHA.119.026240. Epub 2019 Oct 1. PMID 31570084